CLINICAL TRIAL: NCT04977141
Title: Race, Ethnicity, Socioeconomic Status and Prolapse-rElated Decisional ConflicT
Acronym: RESPECT
Status: Completed | Type: Observational
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: Fellows Pelvic Research Network (sponsor) (Unknown); Northwestern University (Other); University of New Mexico (Other); University of California, Irvine (Other); University of South Florida (Other); Emory University (Other); University of Alabama at Birmingham (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Julia Shinnick, MD, Women and Infants Hospital of Rhode Island
Other Study IDs: 1674479
Record Dates: First submitted 2021-07-07; First posted 2021-07-26 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Pelvic Organ Prolapse; Prolapse, Urogenital
Keywords: decisional conflict; pelvic organ prolapse; decision making
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Under-represented minority: Non-English speaking and/or non-White
  Interventions: Other: Decisional Conflict Scale
- Non-under-represented minority: English-speaking and/or White
  Interventions: Other: Decisional Conflict Scale

INTERVENTIONS:
Other: Decisional Conflict Scale — Decisional Conflict Scale

SUMMARY:
This study is trying to see if people from different backgrounds have different feelings when making treatment decisions about prolapse.

DETAILED DESCRIPTION:
This multi-center study will include patients ages >18 years with prolapse symptoms who have new patient consultations to Female Pelvic Medicine and Reconstructive Surgery providers.

After the new-patient consultation, patients will be contacted to see if they are interested in the study. If so, informed consent will be obtained before they complete a 1 page questionnaire that assesses their eligibility for participation.

The questionnaires are: Decisional Conflict Scale; Pelvic Floor Disorders Autonomy Preference Index; Control Preferences Scale; Pelvic Floor Distress Inventory (PFDI 20); Satisfaction with Decision Scale for Pelvic Floor Disorders; Impression questionnaire.

Patients will self-identify their zip-code on the patient impression questionnaire. This will enable a geographic analysis that will assess the relationships of neighborhood and commute on decision making.

For the purposes of this study, patients will self-identify their demographic information.

URM patients will be those who self-identify as having a non-Caucasian race and/or a Hispanic ethnicity. Providers seeing patients that are included in this study will also be consented prior to completing a 1 time demographics questionnaire. Additional clinical data will also be obtained.

Patients will be able to utilize interpreters to participate. Information regarding the use of interpreters will be collected. Questionnaires that are available in, and validated in, non-English languages will be used as appropriate.

The lead study site is Women & Infants Hospital/ Brown University, with additional study sites planning to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Provider inclusion criteria consists of FPMRS providers at study sites seeing new patients with symptoms of pelvic organ prolapse. Patient inclusion criteria consists of new patients 18 years or older with symptoms of pelvic organ prolapse.

Exclusion Criteria:

* Provider exclusion criteria consists of providers who decline participation. Patient exclusion criteria consists of patients who decline participation, and those who cannot complete the study interventions with the assistance of an interpreter.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: New patients with symptoms of pelvic organ prolapse.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Compare Decisional Conflict Scale scores measuring prolapse treatment-related decisional conflict reported by URMs to non-URMs after new patient consultations with FPMRS providers. | immediately on enrollment.

SECONDARY OUTCOMES:
Describe patient and clinical factors associated with increased scores on the Decisional Conflict Scale | immediately on enrollment.
  perform chart review of patient's medical history, self-reported demographic variables, exam findings, symptom scores on the Pelvic Floor Distress Inventory and Decisional Conflict Scale scores
Identify variables correlated with discrepancies between patient-perceived and provider-perceived goals and treatment options | immediately on enrollment.
  Chart review of patient's medical history, exam findings, self-reported demographic variables to investigate if they are correlated with differences in self-reported patient goals and perception of treatment options offered (this is not a named questionnaire, this is a questionnaire developed for the study).
Explore variations in first-line treatments offered and/or selected for pelvic organ prolapse when stratified by race, ethnicity, and socioeconomic status. | immediately on enrollment.
  Chart review of patient's medical history, exam findings, self-reported demographic background to investigate correlation with treatment patterns
Describe a possible correlation between race, ethnicity, and socioeconomic differences with scores on the Patient Autonomy Preferences Index and Patient Control Preferences Scale | immediately on enrollment.
  Review of patient's self-reported demographic background information to assess to correlation with scores on above-mentioned scales.
Describe the association between race, ethnicity, and socioeconomic differences and scores on the Patient Satisfaction with Decision Scale | immediately on enrollment.
  Review of patient's self-reported demographic background information to assess to correlation with scores on above-mentioned scale.
Investigate the relationship between Decisional Conflict Scale scores, Patient Satisfaction with Decision Making scores, and decisional instability 1 year after a new-patient visit. | 1 year
  Review of patient's self-reported demographic background information to assess to correlation with scores on above-mentioned scales.
Investigate a correlation between Decisional Conflict Scale scores and zip-code | immediately on enrollment.
  Review of whether distance driven to a hospital and/or living in a food desert is correlated with a higher Decisional Conflict Scale score.

CONTACTS AND LOCATIONS:
Overall Officials: Julia K Shinnick, MD, Principal Investigator — Women & Infants Hospital
Locations (1):
- Women & Infants Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No